CLINICAL TRIAL: NCT06301204
Title: Evaluation Of The Effectiveness Of Tranexamic Acid Application Protocol With Different Doses On Bleeding, Edema And Physician Comfort In Bimaxillary Orthognathic Surgery Patients
Brief Title: Effectiveness Of Tranexamic Acıd Application Wıth Different Doses On Bleeding, Edema And Physician Comfort In Orthognathıc Surgery Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 21.06.2022-E.67046
Record Dates: First submitted 2024-02-13; First posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Tranexamic Acid; Orthognathic Surgery; Edema; Bleeding
MeSH Terms: conditions — Edema; Hemorrhage | interventions — Tranexamic Acid; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control group (Placebo Comparator): control group patient give no drug administration during bimaxillary orthognathic surgery.
  Interventions: Drug: Saline
- group 1(intravenous administration of 250 mg tranexamic acid) (Active Comparator): group 1 (TRANEXEL 250 mg/5 mL) patients administered 250 mg tnx acid during the whole bimaxillary orthognathic surgery
  Interventions: Drug: Tranexamic acid injection
- group 2 (intravenous administration of 500 mg tranexamic acid) (Active Comparator): group 2 (TRANEXEL 250 mg/5 mL) patients administered 500 mg tnx acid during the whole surgery.
  Interventions: Drug: Tranexamic acid injection

INTERVENTIONS:
Drug: Tranexamic acid injection — tranexamic acid administration 250mg or 500 mg
  Arms: group 1(intravenous administration of 250 mg tranexamic acid); group 2 (intravenous administration of 500 mg tranexamic acid)
Drug: Saline — onyl ıv saline (NaCl 0.09%)
  Arms: control group

SUMMARY:
The aim of this clinical study conducted in accordance with the information in the literature is to compare the effects of administering tranexamic acid during orthognathic surgery, at different doses. Specifically, investigators aim to compare the effects of administering 1 ampoule IV (approximately 3 mg/kg) and 2 ampoules IV (approximately 6 mg/kg), and evaluate their impact on intraoperative bleeding (ml), surgical duration (min), postoperative swelling, and intraoperative surgical field evaluation (Fromme Scale), by comparing them with control group (applying no drug administration) patient data.

DETAILED DESCRIPTION:
This prospective double blind clinical study was approved by the Bezmialem Vakif University Clinical Research Ethics Committee (2022-E.6706). All patients were provided detailed explanations of the surgical procedure and potential adverse events, underwent preoperative anesthesia assessments, and provided informed consent. A total of 60 patients were included in the study and were randomly assigned to three groups: Study Group 1 (N=20), Study Group 2 (N=20), and Control Group (N=20). In Study Group 1, patients received local anesthesia prior to bimaxillary osteotomy, followed by intravenous administration of 250 mg / 2.5 mL tranexamic acid before starting with the incision. In Study Group 2, patients also received local anesthesia before bimaxillary osteotomy, followed by intravenous administration of 250 mg / 2.5 mL tranexamic acid for le fort 1 and, a second dose of 250 mg / 2.5 mL tranexamic acid was administered for beginning of the sagittal split osteotomy. The Control Group, Group 3, did not receive any medication before or after surgery. All patients underwent bimaxillary surgery using the same surgical technique and same surgical team.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with class 2 or class 3 dentofacial malformation who are planned to undergo bimaxillary orthognathic surgery.
2. Patients who have not had orthognathic surgery before
3. Patients without cleft lip and palate
4. Patients without systemic bleeding diets

Exclusion Criteria:

1. Having a systemic disease that affects general health status
2. Presence of a malignant disease in the head and neck region
3. Patients who have previously undergone orthognathic surgery
4. Patients with any bleeding disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
intraoperative bleeding during the surgery (ml) | during the operation time (hour)
  the primary outcome is this study is assessment of the intraoperative bleeding: Intraoperative bleeding will be calculated by subtracting the total amount of iv fluid and the amount of irrigation solutions used during surgery from the total amount of aspirate volume.

SECONDARY OUTCOMES:
postoperative edema calculation for the first 1-3 and 7 day (cm) | post operative 1-3-7 days
  the first secondary outcome of this study is post operative edema: Prior to anesthesia induction, Tragus (Tra) and Gonion (Go) points were marked with methylene blue, and distances including Lateral Canthus - Gonion, Tragus-Commissure, and interincisal distances were measured with a paper ruler and recorded as preoperative measurements.Measurements of Lateral Canthus - Gonion, Tragus-Commissure, and Interincisal distances were repeated on postoperative days 1, 3, and 7 for evaluating postoperative edema.
intraoperative surgical site evaluation (Fromme Scale) | during the surgical time (hour)
  the second secondary outcome is surgical site evaluation during the surgery. Surgeon evaluate the surgical site according to Fromme Scale per every one hour.
  0 = No bleeding, virtually bloodless field
  1. = Bleeding so mild it is not even a surgical nuisance
  2. = Moderate bleeding, a nuisance but without interference with accurate dissection
  3. = Moderate bleeding that moderately compromises surgical dissection
  4. = Heavy but controllable that significantly interferes with dissection
  5. = Massive uncontrollable bleeding
Hemoglobin (Hgb) and Hematocrit (Hct) values alteration preoperative and postoperative 2. day | during the preoperative and post operative 2. day
  Hemoglobin (Hgb) and Hematocrit (Hct) values were recorded preoperatively and second postoperative day.

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakıf Universty, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes